CLINICAL TRIAL: NCT06952153
Title: Comparison of Phaco Surgery and Goniosynechialysis Versus Trabeculectomy Outcomes in Glaucoma Patients
Brief Title: Comparison of Phaco Surgery With Goniosynechialysis Versus Trabeculectomy in Glaucoma Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nguyen Hoang Phuc, Medical Doctor, Principal Investigator, Department of Ophthalmology, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ho Chi Minh City UMP
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Primary Angle Closure Glaucoma
Keywords: PACG; Phaco-GSL; trabeculectomy; RCT; Ophthalmic surgery
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Phacoemulsification; Trabeculectomy; Fluorouracil

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, parallel-group interventional trial. Eligible participants with primary angle-closure glaucoma will be randomly assigned in a 1:1 ratio to undergo either phacoemulsification with goniosynechialysis (Phaco-GSL) or standard trabeculectomy. Randomization will be stratified by baseline age, condition severity and type. All surgical procedures will follow a standardized protocol, and postoperative care will be identical between groups. The primary analysis will compare postoperative intraocular pressure (IOP) and surgical success rates over a 12-month follow-up period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a triple-masked randomized controlled trial with masking of the outcome assessor and data analyst. The surgeon was unmasked due to the nature of surgical interventions, and patients were masked to the study hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard trabeculectomy with 5FU (Active Comparator)
  Interventions: Procedure: Trabeculectomy with 5FU
- Phacoemulsification with Goniosynechialysis (Experimental)
  Interventions: Procedure: Phacoemulsification with Goniosynechialysis

INTERVENTIONS:
Procedure: Phacoemulsification with Goniosynechialysis — This procedure involves standard phacoemulsification cataract surgery combined with goniosynechialysis, which mechanically separates peripheral anterior synechiae to open the anterior chamber angle. It aims to both remove the cataractous lens and restore aqueous outflow in patients with primary angle-closure glaucoma.
  Other Names: Phaco-GSL
  Arms: Phacoemulsification with Goniosynechialysis
Procedure: Trabeculectomy with 5FU — Trabeculectomy is a glaucoma filtration procedure designed to lower intraocular pressure by creating a new drainage pathway from the anterior chamber to the sub-conjunctival space. It is considered the standard surgical intervention for medically uncontrolled glaucoma.
  Arms: standard trabeculectomy with 5FU

SUMMARY:
The goal of this clinical trial is to learn whether phacoemulsification combined with goniosynechialysis (Phaco-GSL) is as effective and safe as trabeculectomy in treating patients with primary angle-closure glaucoma.

The main questions it aims to answer are:

* Does Phaco-GSL provide similar or better intraocular pressure (IOP) control compared to trabeculectomy?
* What are the rates of postoperative complications or adverse events between the two surgical approaches?
* How do the two procedures compare in terms of visual acuity recovery and need for glaucoma medications?

Researchers will compare Phaco-GSL to trabeculectomy to determine which procedure offers better overall outcomes for patients with angle-closure glaucoma.

Participants will:

Be randomly assigned to undergo either Phaco-GSL or trabeculectomy Attend scheduled follow-up visits at regular intervals (e.g., 1 week, 1 month, 3 months, 6 months, 12 months) for eye exams and pressure checks

DETAILED DESCRIPTION:
This clinical trial is designed to compare the clinical efficacy and safety of two surgical interventions for patients with primary angle-closure glaucoma (PACG): (1) phacoemulsification combined with goniosynechialysis (Phaco-GSL), and (2) trabeculectomy. The study is driven by the increasing need to identify surgical approaches that not only provide effective intraocular pressure (IOP) control but also minimize postoperative complications and preserve visual function.

Phacoemulsification with goniosynechialysis aims to address both lens-induced angle crowding and peripheral anterior synechiae (PAS), potentially restoring aqueous outflow through a less invasive approach than trabeculectomy. On the other hand, trabeculectomy remains the gold standard for glaucoma filtration surgery and offers significant IOP reduction, albeit with a higher risk of complications and need for intensive postoperative care.

This randomized, parallel-group, single masked interventional trial will allocate participants to undergo either Phaco-GSL or trabeculectomy. Allocation will be stratified based on key baseline factors age, condition severity and type. All surgical procedures will be performed by experienced glaucoma surgeons following standardized protocols. Postoperative management will be unified across both groups to ensure comparability of outcomes.

Primary and secondary endpoints will include postoperative IOP at predefined intervals, reduction in IOP from baseline, number of anti-glaucoma medications required, visual acuity outcomes, angle status (via gonioscopy), and occurrence of adverse events. Follow-up will extend for at least 12 months to capture both short-term surgical success and medium-term complications or failures.

This trial will provide much-needed data to inform clinical decisions in managing PACG, particularly in cases where lens extraction is indicated. By comparing a combined lens-based and angle-opening procedure to a traditional filtering surgery, the study seeks to clarify the relative benefits and risks of each approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Peripheral anterior synechiae (PAS) >180°
* Glaucomatous optic neuropathy with visual field loss
* Intraocular pressure (IOP) > 21 mmHg despite medication
* Ability to consent and comply with follow-up
* Cataract grade 1 to 3 according to LOCS III
* Best corrected visual acuity (BCVA) ≥ 0.3 logMAR (equivalent to 20/40 Snellen or worse)

Exclusion Criteria:

* Very advanced glaucoma (only light perception vision)
* Secondary angle-closure etiologies
* Prior ocular surgeries or laser peripheral iridotomy (PI)
* Allergy to 5-fluorouracil (5-FU), if used postoperatively
* Irreversible corneal disease
* Chronic corticosteroid use
* Poor follow-up compliance
* Cataract grade 4 or 5 (LOCS III)
* Phacomorphic, phacolytic, or subluxated cataracts

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Mean change in intraocular pressure (IOP) from baseline | 12 months after surgery
  The primary outcome is the mean reduction in intraocular pressure (IOP) measured in mmHg from baseline to the final follow-up visit. IOP will be measured using Goldmann applanation tonometry by a masked outcomes assessor. The purpose is to evaluate the effectiveness of phacoemulsification combined with goniosynechialysis compared to standard trabeculectomy in reducing IOP in patients with primary angle-closure glaucoma.

SECONDARY OUTCOMES:
Change in best-corrected visual acuity (BCVA) from baseline | 12 months postoperatively
  This outcome measures the change in best-corrected visual acuity (BCVA), expressed in logMAR units, from baseline to the final follow-up visit. BCVA will be assessed using standardized ETDRS charts under consistent lighting and testing conditions. The aim is to compare the improvement or decline in visual acuity between participants undergoing phacoemulsification with goniosynechialysis and those undergoing trabeculectomy. Measurements will be conducted by certified examiners masked to group allocation.
Change in number of glaucoma medications from baseline | 12 months postoperatively
  This outcome assesses the difference in the number of topical anti-glaucoma medications used by participants before and after surgery. The total number of medications will be recorded at baseline and at each follow-up visit. The goal is to determine whether phacoemulsification with goniosynechialysis reduces the need for ongoing pharmacological treatment compared to trabeculectomy. A reduction in medication burden is considered an indicator of treatment efficacy and improved patient quality of life.
Change in Total Degree of Angle Closure from Baseline | 12 months postoperatively
  This outcome measure evaluates the change in the extent of angle closure, quantified as the total degrees of the anterior chamber angle that are closed, from baseline to the final follow-up. Assessments will be performed using standardized gonioscopy or anterior segment imaging (e.g., AS-OCT) by examiners masked to treatment allocation. The measurement provides an objective indicator of the anatomical improvement of the angle following intervention, with a reduction in closed angle degrees suggesting a more open drainage pathway, which is critical for effective intraocular pressure control.
Surgical Success Rate | 12 months after surgery
  Surgical success will be classified into two categories:
  Complete Success: Defined by meeting all of the following criteria:
  Postoperative intraocular pressure (IOP) consistently between 5 mmHg and 18 mmHg at each follow-up visit without the use of additional anti-glaucoma medications.
  A ≥20% reduction in IOP from baseline (preoperative value). No need for additional surgical intervention to manage glaucoma. No use of adjunctive glaucoma medications.
  Partial Success: Defined as meeting some but not all criteria for complete success. This may include cases where IOP is within target range but maintained with the aid of medications, or the percentage IOP reduction is less than 20%.
  This outcome provides a comprehensive assessment of surgical effectiveness and will be evaluated at 12 months postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- HCMC University of Medicine and Pharmacy, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the publication (after de-identification) will be shared, including baseline characteristics, intraocular pressure (IOP) values, visual acuity measurements, surgical outcomes, and complication rates. A data dictionary will be provided to facilitate reuse.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the study results and will remain accessible for 2 years.
Access Criteria: Access will be granted to qualified researchers affiliated with academic institutions, non-profit organizations, or healthcare institutions conducting non-commercial research. Requests must include a research proposal and data use agreement. Requests will be reviewed by the study's data access committee.

REFERENCES:
- [Background] Liu Y, Li W, Jiu X, Lei X, Liu L, Yan C, Li X. Systematic Review and Meta-Analysis of Comparing Phacoemulsification Combined with goniosynechialysis to other mainstream procedures in treating patients with angle-closure glaucoma. Medicine (Baltimore). 2019 Oct;98(42):e17654. doi: 10.1097/MD.0000000000017654. PMID 31626152
- [Background] Zhao J, Zhang C, Pazo EE, Dai G, Li Y, Chen Y, Li M, Che H. Phaco-goniosynechialysis versus phaco-trabeculectomy in patients with refractory primary angle-closure glaucoma: a comparative study. BMC Ophthalmol. 2023 Apr 6;23(1):144. doi: 10.1186/s12886-023-02885-6. PMID 37024836